CLINICAL TRIAL: NCT04456725
Title: Intensive Management of At-risk Patients: a Randomized Controlled Trial
Brief Title: Intensive Management of At-risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CareMore Health, San Bernardino (Other)
Responsible Party: Principal Investigator, Paul Bixenstine, Primary Care Physician, CareMore Health, San Bernardino
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-06-21; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Chronic Disease
Keywords: high need high cost; population health; care management; quality improvement; ambulatory care; primary care; readmission prevention
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be informed that their care is different than usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Usual care group
  Interventions: Behavioral: Control
- Intervention (Experimental): Intensive management utilizing longitudinal patient tracking, proactive outreach, multidisciplinary action planning and careful outcomes monitoring.
  Interventions: Behavioral: Intensive management

INTERVENTIONS:
Behavioral: Intensive management — The intervention group will be assigned to a partnership of one nurse practitioner and one medical assistant who will manage them intensively, with the support of the study team.
  Arms: Intervention
Behavioral: Control — Usual care
  Arms: Control

SUMMARY:
The purpose of this study is to assess if intensive management of at-risk participants, utilizing longitudinal patient tracking, proactive outreach, multidisciplinary action planning and careful outcomes monitoring, will lead to better patient outcomes than usual care.

DETAILED DESCRIPTION:
At-risk participants will be randomized 1:1 to either usual care or intensive management utilizing longitudinal patient tracking, proactive outreach, multidisciplinary action planning and careful outcomes monitoring for 6 months. Participants in the intervention group will be assigned to a partnership of one nurse practitioner and one medical assistant who will manage them with the support of the study team. Staff will focus on contacting all patients within one week of any emergency department visit or hospital discharge, contacting all highest-risk participants weekly and all participants monthly, and completing high-priority tasks for participant care within one week. The primary outcomes of this quality improvement study are inpatient bed days and number of inpatient admissions.

ELIGIBILITY:
Inclusion Criteria: At-risk patients, meaning Gold, Silver, or Bronze tier, as identified by our member 360 platform:

* Gold tier - 6+ emergency department (ED) visits last year, annual spend >$100,000, 8 or more hierarchical condition category (HCC) diagnoses, readmission <30 days prior, or ambulatory care-sensitive condition (ACSC) hospitalization <30 days prior
* Silver tier - 4+ ED visits last year, annual spend >$75,000, 6 or more HCC diagnoses, readmission <90 days prior, substance abuse HCC diagnosis, behavioral health admit <90 days, 15+ chronic medications prescribed in the last 90 days (and not qualifying for Gold tier)
* Bronze tier - 3+ ED visits last year, annual spend >$50,000, 5 or more HCC diagnoses, 3+ hospitalizations last year, end-stage liver disease, end-stage renal disease, Medicare and Medicaid dual-enrolled, disease-management program patients with ACSC admission or ED visit in the last year, 10+ chronic medications in the last 90 days, 6+ health risk-assessment score, 12+ Edmonton Frail Scale score (and not qualifying for Gold or Silver tiers)

Exclusion Criteria:

* enrolled in hospice
* enrolled in Institutional Special Needs Plan
* primary patient of study investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
inpatient bed days | 6 months
  number of total participants' days of care in an inpatient setting
inpatient admissions | 6 months
  total number of participants' inpatient admissions

SECONDARY OUTCOMES:
ED visits | 6 months
  participants' total emergency department visits
30-day readmissions | 30 days
  participants' total inpatient readmissions within 30 days
180-day readmissions | 180 days
  participants' total inpatient readmissions within 180 days
ACSC admits | 6 months
  participants' inpatient admissions for ambulatory care sensitive conditions
inpatient plus SNF bed days | 6 months
  number of total days of participants' care in an inpatient or skilled nursing facility setting
cost | 6 months
  participants' total medical expenditures
delta MLR | 6 months
  average change in each participant's medical loss ratio
average percent post-acute contact within 1 week | 1 week
  average percent of participants contacted within 1 week of emergency department visit, hospital or skilled-nursing facility discharge
average percent of high-priority tasks completed within 1 week | 1 week
  average percent of participant care tasks designated as high-priority that are completed within 1 week of being assigned
average percent of Gold patients contacted weekly | 1 week
  average percent of participants in Gold tier contacted every week
average percent of participants contacted monthly | 1 month
  average percent of participants contacted every 4 weeks
average change in percent of high-priority HEDIS gaps | 6 months
  average change in percent of open Healthcare Effectiveness Data and Information Set (HEDIS) measures that are high-priority, meaning statin use in diabetics and cardiovascular disease; medication adherence for oral diabetes, hypertension and statin; diabetes A1c control; and blood pressure control
average change in staff satisfaction score | 6 months
  average difference in sum of Likert scale responses to staff satisfaction survey
average change in participant satisfaction score | 6 months
  average difference in sum of Likert scale responses to participant satisfaction survey

OTHER OUTCOMES:
average change in RAF | 6 months
  average change in each participant's Risk Adjustment Factor
average number of high-priority tasks completed per week | 1 week
  average number of participant care tasks designated high-priority completed per week
average time on high-priority tasks per week | 1 week
  average amount of time in minutes per week spent by staff in attempting to complete high-priority participant care tasks
number of in-person visits | 6 months
  total number of in-person care visits by participants

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bixenstine, MD, Principal Investigator — CareMore Health

IPD SHARING:
Plan to Share IPD: No